CLINICAL TRIAL: NCT05644964
Title: The Effect of Anemia in Adolescent and Advanced Age Pregnancies on the Tissue of the Placenta
Brief Title: The Effect of Anemia in Adolescent and Advanced Age Pregnancies
Status: Completed | Type: Observational
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Hayrunnisa Yesil Sarsmaz, Asistant Prof., Celal Bayar University
Other Study IDs: MCBU_anemia
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Anemia Pregnancy; Placenta Diseases
Keywords: anemia in pregrnancy; Placenta; Risky Pregnancy; immunohistochemistry; Aging
MeSH Terms: conditions — Placenta Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — placenta tissues
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1:: Anemic pregnancies under the age of 18 (study group),
- Group 2:: Anemic pregnancies over the age of 35 (study group)
- Group 3:: Pregnant women under the age of 18 are not anemic (control group)
- Group 4:: Non-anemic pregnant women over the age of 35 (control group)

SUMMARY:
Anemia by the Centers for Disease Control and Prevention (CDC, 1989); It is defined as hemoglobin (Hb) or

hematocrit (Hct) values below the 5th percentile in pregnant women. It is expressed as Hb value of 11 mg / dl

or Hct value below 33% in the first trimester. II. Less than 10.5 g / dl in trimester can be defined as anemia.

Anemia is a risk factor during pregnancy and one of the predisposing causes of maternal death. Pregnancy

anemia can be aggravated by various conditions such as uterine or placental bleeding, gastrointestinal

bleeding and peripartum blood loss. In addition to the general consequences of anemia, there are specific risks for the mother and fetus during pregnancy such as intrauterine growth retardation, prematurity, feto-placental miss rate, and higher risk for peripartum blood transfusion. Literature studies on anemia in risky age groups during pregnancy (adolescence and advanced age pregnancy) have been reviewed. Some articles and theses published in Turkey and abroad were found. However, the number of studies related to the study subject in Turkey is quite small. For this reason, conducting a research on the effect of anemia on the placenta during pregnancy will lead to a decrease in the gap in the literature and an increase in the awareness of the public on the subject when the research results are obtained. The research is of a prospective type. The universe of the study will be composed of pregnant women who voluntarily agree to participate in the study chosen by the improbable sampling method. According to the anemia of the pregnant women within the scope of the research; I: Group: Anemic pregnancies under the age of 18 (study group), II: Group: Anemic pregnancies over the age of 35 (study group) III: Group : Pregnant women under the age of 18 are not anemic (control group) IV: Group : Non-anemic pregnant women over the age of 35 (control group) as planned. The placentas of pregnant women who gave birth between 37-42 weeks of age and who voluntarily accepted to participate in the study and who were compatible with age and parity will be examined histopathologically, with a total of at least 30 placentas from each group. Those who had an out-of-term delivery, had multiple pregnancy, preeclampsia, gestational diabetes mellitus, thyroid dysfunction, systemic diseases other than anemia, and those who used drugs other than anemia during pregnancy will not be included in the study. The research will only be conducted with women who have a normal vaginal delivery. In our research, it will be examined whether the possible changes that anemia (anemia) will make in the expression of IRP protein 1 produced from the placenta affect the placenta and the baby. In addition, the relationship between IRP protein 1 and primary related TFrP 1 and indirectly changes in DMT1 expressions will be evaluated, so that the intrauterine growth retardation (IUGG), which is one of the negative effects of anemia in pregnancy, and TFrP 1, are the molecules that increase the end-stage release from the placenta. and its relationship in terms of Dmt1 molecules will be investigated. The tissue samples of placenta that will be obtained after the experiment periods, will be buried in paraffin-embedded blocks after routine tissue tracing, and from the obtained blocks, 5 microns of incisions will be taken via microtome, which will then be stained with Hematoxylin-Eosin and then HPL, IGF and leptin expression levels will be examined with the light microscope by immunohistochemical staining. The results of the research data created by determining the effect of the histopathological examinations on the placentas of women with anemia seen in pregnant women in risky age groups will be a source for the next studies. Maternal anemia (of the mother) seen in pregnancies has been studied many times before, but maternal anemia seen in adolescents and advanced age groups will add a different dimension to the subject and will shed light on other studies on the subject. In this way, it is aimed to draw attention to other researches to be carried out to take the necessary measures and measures against these problems.

ELIGIBILITY:
Inclusion Criteria:

* Clinic diagnosis of anemic pregnancies
* Pregnant women who have spontaneous vaginal birth
* Anemia in Adolescent Pregnancy
* Anemia in Advanced Age Pregnancy

Exclusion Criteria:

* multiple pregnancy
* insulin dependent diabetes
* pregnant women who have had a cesarean section
* preeclampsia
* thyroid disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: anemic pregnant women under the age of 18, Anemic pregnant women over the age of 35, not anemic pregnant women under age of 18 and not anemic pregnant women over the age of 35
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
%22,2 Patients's placenta with Anemia in Adolescent ( ≤18)Pregnancy and %26,7 Patients's Placenta with from Anemia in Advanced Age (≥35) Pregnancy. Placenta Tissues Staining Measured by immunohistochemistry tecnique. | Baseline
  DMT1, TFR1 and IRP1 immunohistochemistry results are higher in anemic pregnants compared to non-anemic pregnant women aged ≤18 and ≥35 years. Even if the mother has iron deficiency, the deficiency can be tolerated by the iron absorption mechanism in the placenta.

CONTACTS AND LOCATIONS:
Overall Officials: Ada Israfilzade, Researcher asist, Study Chair — Manisa Celal Bayar University; Gulsen Gurgen, Assoc.Dr., Study Chair — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University, Yunusemre, Mani̇sa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes